CLINICAL TRIAL: NCT03916289
Title: Establishing A National Tiered Diagnosis and Treatment System of Osteoporosis in China: A Pilot Study
Brief Title: A Tiered Management System of Osteoporosis in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS-1894
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Osteoporosis; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention would be taken — No intervention would be taken. Patients enrolled would be managed by this tiered diagnosis and treatment system and receive standard treatment according to clinical guidelines of osteoporosis.

SUMMARY:
There is a management gap in China. This study aims to establish a tiered management system of osteoporosis for Chinese patients. Including:

1. Developing a national hierarchical health management network platform for middle-aged and elderly osteoporosis patients. With this platform, the data of medical records, laboratory results would be shared between medical institutions. And primary hospitals can refer the patients to the nearest medical centre for advanced auxiliary examinations and diagnosis.
2. Establishing a muti-level hospital collaboration, doctor-patient interaction management model of osteoporosis.
3. To explore and establish a early warning and screening pathways for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women or men aged 50 years or older

Conform to the diagnosis of osteoporosis or osteopenia as followings:

1. Bone mineral density measured by dual-energy X-ray absorptiometry show a T-score ≤ -1.0 at neck of femur or total hip or lumber 1-4 OR
2. Have at least once major osteoporotic fracture

Exclusion Criteria:

* Screened people who do not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community population and outpatients in each clincal centre
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled at year 1 | Year 1
  The number of patients with osteoporosis or osteopenia enrolled in each medical centre at year 1
Number of patients enrolled at year 2 | Year 2
  The number of patients with osteoporosis or osteopenia enrolled in each medical centre at year 2
Number of patients enrolled at year 3 | Year 3
  The number of patients with osteoporosis or osteopenia enrolled in each medical centre at year 3

SECONDARY OUTCOMES:
Number of patients screened at year 1 | Year 1
  The number of patients screened for osteoporosis in each medical centre at year 1
Number of patients screened at year 2 | Year 2
  The number of patients screened for osteoporosis in each medical centre at year 2
Number of patients screened at year 3 | Year 3
  The number of patients screened for osteoporosis in each medical centre at year 3
The proportion of patients treated in compliance with guidelines at year 1 | Year 1
  The proportion of patients treated in compliance with guidelines at year 1
The proportion of patients treated in compliance with guidelines at year 2 | Year 2
  The proportion of patients treated in compliance with guidelines at year 2
The proportion of patients treated in compliance with guidelines at year 3 | Year 3
  The proportion of patients treated in compliance with guidelines at year 3
Data integrity in network platform at year 1 | Year 1
  The integrity of data recorded in network platform. Including general characteristics (name, sex, age, height, weight and race), medical history (onset age, chief complaint, history of fractures, medication history, previous history and family history), results of auxiliary examinations (DXEA is mandatory required, and other examinations may differ between medical centres, usually including serum calcium, serum phosphorus, serum total alkaline phosphatase, urine calcium, urine phosphorus, serum parathyroid hormone, X ray of vertebrae and so on), prescriptions, and follow-up data. At year 1.
Data integrity in network platform at year 2 | Year 2
  The integrity of data recorded in network platform. Including general characteristics (name, sex, age, height, weight and race), medical history (onset age, chief complaint, history of fractures, medication history, previous history and family history), results of auxiliary examinations (DXEA is mandatory required, and other examinations may differ between medical centres, usually including serum calcium, serum phosphorus, serum total alkaline phosphatase, urine calcium, urine phosphorus, serum parathyroid hormone, X ray of vertebrae and so on), prescriptions, and follow-up data. At year 2.
Data integrity in network platform at year 3 | Year 3
  The integrity of data recorded in network platform. Including general characteristics (name, sex, age, height, weight and race), medical history (onset age, chief complaint, history of fractures, medication history, previous history and family history), results of auxiliary examinations (DXEA is mandatory required, and other examinations may differ between medical centres, usually including serum calcium, serum phosphorus, serum total alkaline phosphatase, urine calcium, urine phosphorus, serum parathyroid hormone, X ray of vertebrae and so on), prescriptions, and follow-up data. At year 3.

CONTACTS AND LOCATIONS:
Overall Officials: The propotion of patients treated in comliance with guidelines Xia, MD, Study Chair — Peking Union Medical College Hospital
Locations (25):
- China (25):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing shijingshan hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The third hospital of hebei medical university, Shijiazhuang, Hebei
  - The Second Hospital of Xiangya,Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The fourth hospital of jilin university, Changchun, Jilin
  - Shengjing hospital affiliated to China medical university, Shenyang, Liaoning
  - People's hospital of ningxia hui autonomous region, Yinchuan, Ninxia
  - The Sixth People's Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Huadong hospital affiliated to fudan university, Shanghai, Shanghai Municipality
  - Shanghai first people's hospital affiliated to Shanghai jiaotong university, Shanghai, Shanghai Municipality
  - Tongji hospital affiliated to tongji university, Shanghai, Shanghai Municipality
  - Xi'an Red Cross hospital, Xi'an, Shannxi
  - The first affiliated hospital of shanxi medical university, Taiyuan, Shanxi
  - West China hospital of sichuan university, Chengdu, Sichuan
  - Western theater general hospital, Chengdu, Sichuan
  - Tianjin hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No